CLINICAL TRIAL: NCT02506439
Title: Randomized Controlled Trial to Determine the Nutritional Requirement for Vitamin D for Prevention of Deficiency During Pregnancy and in the Early Neonatal Period (D-MAT)
Brief Title: Nutritional Requirements for Vitamin D in Pregnant Women
Acronym: DMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Mairead Kiely PhD, Professor of Human Nutrition, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ODINWP4DMAT
Record Dates: First submitted 2015-05-12; First posted 2015-07-23 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Cholecalciferol; Dose-response; Randomized Controlled Trial; Pregnancy; Cord blood; Serum 25-hydroxyvitamin D; Vitamin D Deficiency; Nutrition; Dietary intervention study
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- 10 mcg Vitamin D3 (Experimental): White-skinned women will receive Cholecalciferol (Vitamin D3) 10 mcg [400 IU] daily
  Interventions: Dietary Supplement: 10 mcg Vitamin D3
- 20 mcg Vitamin D3 (Experimental): White-skinned women will receive Cholecalciferol (Vitamin D3) 20 mcg [800 IU] daily
  Interventions: Dietary Supplement: 20 mcg Vitamin D3
- Placebo (Placebo Comparator): White-skinned women will receive a Placebo supplement, identical in appearance and taste to the active product
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 10 mcg Vitamin D3 — Once daily, 10mcg (400IU) dose of vitamin D3 taken from baseline visit (approx 15 weeks gestation) until endpoint (delivery)
  Other Names: Cholecalciferol
  Arms: 10 mcg Vitamin D3
Dietary Supplement: 20 mcg Vitamin D3 — Once daily, 20mcg (800IU) dose of vitamin D3 taken from baseline visit (approx 15 weeks gestation) until endpoint (delivery)
  Other Names: Cholecalciferol
  Arms: 20 mcg Vitamin D3
Dietary Supplement: Placebo — Once daily, placebo capsule containing 0mcg (0IU) of vitamin D3 taken from baseline visit (approx 15 weeks gestation) until endpoint (delivery)
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
Randomised, placebo-controlled dose-response intervention study with vitamin D3 in pregnant women.

DETAILED DESCRIPTION:
This is a three-arm, parallel, double-blind, placebo-controlled dose-response intervention study with vitamin D3. Women will be recruited prior to 18 weeks of gestation and randomised to receive placebo, 10 or 20 mcg/d of vitamin D3 from baseline visit in their first trimester until delivery. Blood samples will be collected at baseline, midpoint and endpoint of the trial, at 10 week intervals, and from the umbilical cord at delivery. A 25-hydroxyvitamin D concentration of 30 nmol/L will be used to denote vitamin D deficiency. Information on maternal anthropometry, diet, lifestyle, sun exposure, blood pressure, iPTH and serum total calcium will also be reported.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* No more than 18 weeks gestation
* In good general health
* Low risk pregnancy
* Not consuming >10 mcg/d vitamin D from supplements

Exclusion Criteria:

* Current smokers
* Diagnosed hypertension
* Known high-risk pregnancy
* Diagnosed medical illness including diabetes mellitus (Types 1 & 2), chronic kidney disease or gastro-intestinal diseases or any illness known to interfere with calcium metabolism (e.g. sarcoidosis).
* Consumption of medications known to interfere with vitamin D metabolism
* Consumption of vitamin D (≥ 10 µg/day) or calcium (≥ 650 mg/d) supplements prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D in pregnant women and cord blood | Change from 1st through 2nd trimester and at delivery
  Analysis of serum 25-hydroxyvitamin D in mothers for blood taken in the first, second and third trimesters and in umbilical cord

SECONDARY OUTCOMES:
Serum total calcium | Change from 1st through 2nd trimester and at delivery
  Analysis of serum total calcium (adjusted for albumin) in mothers for blood taken in the first, second and third trimesters and in umbilical cord
Serum Parathyroid Hormone | Change from 1st through 2nd trimester and at delivery
  Analysis of serum PTH in mothers for blood taken in the first, second and third trimesters and in umbilical cord

CONTACTS AND LOCATIONS:
Overall Officials: Mairead Kiely, PhD, Principal Investigator — University College Cork
Locations (2):
- Ireland (2):
  - Cork University Maternity Hospital and University College Cork, Cork
  - Human Nutrition Resource Unit, School of Food and Nutritional Sciences, University College Cork, Cork

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be considered, for vitamin D intake and 25(OH)D data. Please contact m.kiely@ucc.ie.

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] O'Callaghan KM, Hennessy A, Hull GLJ, Healy K, Ritz C, Kenny LC, Cashman KD, Kiely ME. Estimation of the maternal vitamin D intake that maintains circulating 25-hydroxyvitamin D in late gestation at a concentration sufficient to keep umbilical cord sera >/=25-30 nmol/L: a dose-response, double-blind, randomized placebo-controlled trial in pregnant women at northern latitude. Am J Clin Nutr. 2018 Jul 1;108(1):77-91. doi: 10.1093/ajcn/nqy064. PMID 29878035